CLINICAL TRIAL: NCT02646774
Title: A Multi-center, Open-label, Non-comparative Study to Evaluate the Efficacy and Safety of Micafungin Against Invasive Aspergillosis (CFDA Commitment)
Brief Title: Post Marketing Study to Evaluate the Efficacy and Safety of Micafungin Treatment on Invasive Aspergillosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to administrative reasons
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACN-MA-MYC-IA-2012
Record Dates: First submitted 2015-12-16; First posted 2016-01-06 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Invasive Aspergillosis
Keywords: Aspergillosis; Antifungal; Micafungin
MeSH Terms: conditions — Aspergillosis | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micafungin group (Experimental): Injection
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Injection

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of intravenous micafungin for the treatment of proven or probable fungal infections caused by Aspergillus sp. (Fungemia, respiratory mycosis, gastrointestinal mycosis) in adult patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as proven or probable infections caused by aspergillus (including fungemia, respiratory mycosis and gastrointestinal mycosis) with reference to the definition of EORTC/MSG
* Females of childbearing potential are not pregnant in the study and reliable methods of contraception should be maintained during the whole study.
* Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study is obtained.

Exclusion Criteria:

* Patient received any echinocandins drug within 1 month prior to enrollment.
* Patient was enrolled in any other clinical study within the last month.
* AST/ALT > 5 times the upper limit of normal (ULN)
* total bilirubin> 2.5 times ULN
* BUN/Ccr > 3 times ULN
* HIV positive patient
* Patient has a history of hypersensitivity, or any serious reaction to any component of this product or other echinocandins.
* Patient has a life expectancy of <1 month
* Subject is unlikely to comply with the visits scheduled in the protocol in the opinion of investigator or has a history of non-compliance.
* Pregnant women, nursing mothers, lactating women, and women of child-bearing potential who are unwilling to use reliable contraception for the duration of the study and for 6 weeks following completion of the study.
* Patient has been previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-06-26 (Actual); Study Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
Overall success rate for patients with no hematology disease | At the end of the treatment (up to a maximum of 4 weeks)
  Overall success rate = number of success patients/number of patients for efficacy evaluation x 100% at end of treatment (overall success is defined as patients with complete or partial response)
Overall success rate for patients with hematology disease | At the end of the treatment (up to a maximum of 12 weeks)
  Overall success rate = number of success patients/number of patients for efficacy evaluation x 100% at end of treatment (overall success is defined as patients with complete or partial response)

SECONDARY OUTCOMES:
Clinical improvement rate for patients with no hematology disease | Week 1 up to the end of the treatment (up to a maximum of 4 weeks)
Clinical Improvement rate for patients with hematology disease | Week 1 up to the end of the treatment (up to a maximum of 12 weeks)
Fungal clearance rate for patients with no hematology disease | Week 1 up to the end of the treatment (up to a maximum of 4 weeks)
Fungal clearance rate for patients with hematology disease | Week 1 up to the end of the treatment (up to a maximum of 12 weeks)
Fatality rate for patients with no hematology disease | End of the treatment (up to 2 weeks, and up to 4 weeks for refractory patients)
Fatality rate for patients with hematology disease | End of the treatment (up to 6 weeks, and up to 12 weeks for refractory patients)
Percentage of participants with common Aspergillus infection sites | End of treatment (up to 12 weeks)
Safety assessed by adverse events | Up to 2 weeks after end of treatment (up to14 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (19):
- China (19):
  - Beijing
  - Changsha
  - Chengdu
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Harbin
  - Hefei
  - Hengyang
  - Jinan
  - Nanchan
  - Shanghai
  - Shijiazhuang
  - Suzhou
  - Taiyuan
  - Tianjing
  - Wenzhou
  - Wuhan
  - Zhengzhou

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=167